## **Informed Consent.**

**Study Title**: Role OF OCT-A TO Detect Possible Retinal Vascular Complications of Sofosbuvir (Sovaldi) in Patients With Hepatitis C Virus Infection

Principle Investigators: Prof. Dr. Magda SalahEldin

Date: //

You are invited to participate in a research study conducted by Mohamed Saad from the faculty of medicine, Cairo University. We are asking you to take part in this study to prospectively evaluate the value of Optical coherence tomography angiography (OCT-A) for the of detection of suspected retinal complications With Sofosbuvir (Sovaldi) in Patients With Hepatitis C Virus Infection.

Your participation is voluntary and would consist of comprehensive ophthalmic examination including: Manifest refraction ,Corrected distance visual acuity ,Anterior segment examination using slit lamp and tear film breakup time test, Fundus examination and Recent Optical coherence tomography angiography (OCT-A) will be performed before Treatment Administration and after finishing Course.

There are no anticipated risks to your participation and there are no direct benefits to you for taking part in this study.

You will receive a free ophthalmic examination and follow during period of treatment course for your participation. You will be given a copy of this form.

If you have any questions about this research study, please contact: +201007654385.

| If you | agree fo | or participati | on please | sign here | : | • |
|---|---|---|---|---|---|---|